CLINICAL TRIAL: NCT02541942
Title: Pharmacogenetic Testing of Saliva Samples From Patients With Five or More Exposure Days to rFVIIa Analogue in the Adept 2 Trial
Brief Title: Pharmacogenetic Testing of Saliva Samples From Patients With Five or More Exposure Days to rFVIIa Analogue in the Adept™2 Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NN1731-4214; 2015-001919-13 (EudraCT Number); U1111-1169-6103 (Other: WHO)
Record Dates: First submitted 2015-08-19; First posted 2015-09-04 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collection of specimen (Other)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — For patient convenience, genetic material will be collected in the form of saliva samples.

SUMMARY:
This study is conducted globally. This study describes pharmacogenetic testing of saliva samples from patients who participated in the NN1731-3562 trial (adept™2) (NCT01392547). The objective is to determine the HLA (human leukocyte antigen) type and polymorphisms in the FVII gene in patients previously exposed to rFVIIa analogue.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before collection of saliva samples
* Previous participation in adept™2 trial with 5 or more exposure days to rFVIIa analogue

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- United States (5):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Boston, Massachusetts
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Japan (3):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Timișoara, Timiș County, Romania
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Novi Sad
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 16 sites in 7 countries, as follows: Greece: 2 sites; Japan: 3 sites; Malaysia: 1 site, Romania 1 site, Serbia: 2 sites; Thailand: 2 sites; United States: 5 sites.
Pre-assignment Details: This trial describes pharmacogenetic testing of saliva samples from patients who participated in the completed NN1731-3562 (adeptTM2) phase 3 trial, with 5 or more exposure days to trial product rFVIIa analogue.
Groups:
- Subjects for Analysis: Patients who participated in the completed NN1731-3562 (adeptTM2) phase 3 trial, with 5 or more exposure days to trial product rFVIIa analogue and/or rFVIIa, were included in this arm.
Period: Overall Study
Arm/Group | Subjects for Analysis
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects for Analysis
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — This table reflects the age of the patients when entering the preceding main triall NN1731-3562.
  years | 25.26 (11.69)
Age, Customized [Number; unit: Participants] — This table reflects the age of the patients when entering the preceding main trial NN1731-3562.
  Participants
    Adolescents (12-17 years) | 4
    Adults (18-64 years) | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Determination of HLA Type
Description: HLA typing includes up to 8 different HLA types (HLA-DRB1/B3/B4/B5, DPA1/B1 and DQA1/B1) and their most likely alleles. Number of participants with most likely HLA allele are reported.
Time Frame: Up to 12 months
Population: All enrolled patients
Measure: Number; unit: subjects
Arm/Group | Subjects for Analysis
Number analyzed (Participants) | 19
subjects
  HLA-DPA1*01:03 | 15
  HLA-DPA1*02:01 | 5
  HLA-DPA1*02:02 | 5
  HLA-DPB1*01:01 | 1
  HLA-DPB1*02:01 | 1
  HLA-DPB1*03:01 | 3
  HLA-DPB1*04:01 | 11
  HLA-DPB1*04:02 | 6
  HLA-DPB1*05:01 | 4
  HLA-DPB1*09:01 | 1
  HLA-DPB1*11:01 | 1
  HLA-DPB1*13:01 | 2
  HLA-DPB1*14:01 | 1
  HLA-DPB1*17:01 | 1
  HLA-DPB1*23:01 | 1
  HLA-DQA1*01:01 | 8
  HLA-DQA1*01:02 | 5
  HLA-DQA1*01:03 | 3
  HLA-DQA1*02:01 | 1
  HLA-DQA1*03:01 | 6
  HLA-DQA1*04:01 | 1
  HLA-DQA1*05:01 | 7
  HLA-DQB1*02:01 | 3
  HLA-DQB1*02:02 | 1
  HLA-DQB1*03:01 | 4
  HLA-DQB1*03:02 | 3
  HLA-DQB1*03:03 | 1
  HLA-DQB1*04:01 | 2
  HLA-DQB1*04:02 | 2
  HLA-DQB1*05:01 | 7
  HLA-DQB1*05:02 | 2
  HLA-DQB1*05:03 | 1
  HLA-DQB1*06:02 | 2
  HLA-DQB1*06:03 | 3
  HLA-DQB1*06:04 | 1
  HLA-DQB1*06:09 | 1
  HLA-DRB1*01:01 | 3
  HLA-DRB1*01:02 | 1
  HLA-DRB1*03:01 | 3
  HLA-DRB1*04:03 | 1
  HLA-DRB1*04:04 | 2
  HLA-DRB1*04:05 | 2
  HLA-DRB1*07:01 | 1
  HLA-DRB1*08:02 | 1
  HLA-DRB1*08:04 | 1
  HLA-DRB1*09:01 | 1
  HLA-DRB1*10:01 | 2
  HLA-DRB1*11:01 | 2
  HLA-DRB1*11:04 | 2
  HLA-DRB1*13:01 | 3
  HLA-DRB1*13:02 | 2
  HLA-DRB1*13:05 | 1
  HLA-DRB1*14:01 | 2
  HLA-DRB1*15:01 | 2
  HLA-DRB1*15:02 | 2
  HLA-DRB1*16:01 | 1
  HLA-DRB3*01:01 | 5
  HLA-DRB3*02:02 | 5
  HLA-DRB3*03:01 | 2
  HLA-DRB4*01:01 | 5
  HLA-DRB5*01:01 | 2
  HLA-DRB5*01:02 | 2
  HLA-DRB5*02:02 | 1

2. Primary Outcome: Determination of Polymorphisms in the FVII Gene
Description: Determination of polymorphisms in the FVII gene in patients who participated in the completed NN1731-3562 (adeptTM2) phase 3 trial, with 5 or more exposure days to trial product rFVIIa analogue and/or rFVIIa.
Time Frame: Up to 12 months
Measure: Number; unit: Number of polymorphism
Arm/Group | Subjects for Analysis
Number analyzed (Participants) | 19
Number of polymorphism | 0

ADVERSE EVENTS:
Description: This is a bio-specimen research study. There is no safety data collected and no analysis done in this trial.
Arm/Group | Subjects for Analysis
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.